CLINICAL TRIAL: NCT03910868
Title: Study of the Impact of P-gp, MRP2, ENT-1 and CNT3 on the Blood Concentration / Intra-PBMC Concentration of Tacrolimus in Liver and Kidney Transplant Patients
Brief Title: Impact of P-gp, MRP2, ENT-1 and CNT3 on the Blood Concentration / Intra-PBMC Concentration of Tacrolimus
Acronym: TRANS-TAC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30018_TRANS-TAC
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Liver Transplantation; Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective and monocentric pharmacokinetic study

DETAILED DESCRIPTION:
Membrane transporters supporting tacrolimus at the lymphocyte level may play a role in the variability of the relationship between tacrolimus blood concentration and intracellular concentration, or may be the main explanatory factors. Nevertheless, most of the studies carried out on the subject, have been by genetic approach, neglecting in fact the membrane expression of these transporters, which could testify more to the real effect on the transport of tacrolimus. A better understanding of the cellular transport mechanisms of tacrolimus in the T lymphocyte could thus make it possible to identify sub-populations of patients under-exposed at the intra-lymphocyte level, despite satisfactory systemic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adult of 18 or over;
* fully and honestly informed, and not having reported his non-opposition to the use of his samples for research;
* Affiliated to a social security scheme;
* Hepatic and / or renal transplant stable between two and twenty-four months after transplantation, treated with tacrolimus;
* Without modification of immunosuppressive treatment or treatment likely to modify their pharmacokinetics (imidazoles, macrolides ...) during the last two weeks;
* Each patient can only be included once.

Exclusion Criteria:

* Participation in another protocol whose procedures are incompatible with the realization of the study;
* Pregnant woman ;
* Major person subject to legal protection (safeguard of justice, guardianship, tutorship);
* Person deprived of liberty;
* Opposition to the use of clinical data and remnants of samples taken from care for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatic and / or renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Correlation between drug transporters expression (RNA and protein) in PBMC and tacrolimus intra-PBMC concentration | During the consultation (between 2 and 24 months after the transplant)
  The mRNA levels will be recorded as a cycle threshold difference between the studied gene, and the mean of two housekeeping genes (ACTB and B2M). The proteic expression of the studied transporters will be recorded as fluorescent intensity levels

SECONDARY OUTCOMES:
Correlation between drug transporters RNA expression in PBMC and drug transporters protein expression in PBMC | During the consultation (between 2 and 24 months after the transplant)
  The mRNA levels will be recorded as a cycle threshold difference between the studied gene, and the mean of two housekeeping genes (ACTB and B2M). The proteic expression of the studied transporters will be recorded as fluorescent intensity levels
Correlation between tacrolimus blood to intracellular ratio and adverse events. | During the consultation (between 2 and 24 months after the transplant)
  Tacrolimus-related adverse effects as recorded on the medical record of the patient.
Correlation between tacrolimus intra-PBMC concentration and treatment outcome | During the consultation (between 2 and 24 months after the transplant)
  Treatment outcome as recorded on the medical record of the patient.
Correlation between tacrolimus intra-PBMC concentration and comedications | During the consultation (between 2 and 24 months after the transplant)
  Co-medications as recorded on the medical record of the patient.
Correlation between tacrolimus intra-PBMC concentrations and Donor Graft cell-free DNA (cf-DNA) concentration | During the consultation (between 2 and 24 months after the transplant)
  Donor graft cf-DNA characterized the cell death marker, released from necrotic or apoptotic cells in the transplant organ, and may therefore be useful as a marker for graft injury. When its plasma concentration increases, it evidences that a lesion process occurs in the graft

CONTACTS AND LOCATIONS:
Overall Officials: Florian LEMAITRE, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France